CLINICAL TRIAL: NCT03411512
Title: Tissue Oxygenation in Newborns With Congenital Heart Defects
Brief Title: Congenital Heart Defects and NIRS
Status: Completed | Type: Observational
Sponsor: Petja Fister, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Petja Fister, MD, PhD, Principal Investigator, Petja Fister, MD, PhD, University Medical Centre Ljubljana
Organization: University Medical Centre Ljubljana (Other)
Other Study IDs: NIRS CHD1
Record Dates: First submitted 2018-01-19; First posted 2018-01-26 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Heart Defects, Congenital
Keywords: congenital heart defects; near-infrared spectroscopy; newborn; tissue oxygenation
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CHD: Newborns with structural congenital heart defects. The exclusion criteria were pulmonary or neurological disease, perinatal asphyxia, acute illness, prematurity and congenital abnormality other than CHD.
- Healthy controls: The control group comprised of healthy matched newborns without a diagnosed CHD.

SUMMARY:
Congenital Heart Defects and NIRS

DETAILED DESCRIPTION:
Brain, kidney and intestinal tissue oxygenation in newborns with congenital heart defects assessed by near-infrared spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

Investigators included term newborns with critical structural CHD (of different types) who required surgical or transcatheter procedure in the first year of life. CHD were diagnosed by pediatric cardiologist by clinical examination and echocardiography.

Exclusion Criteria:

The exclusion criteria were pulmonary or neurological disease, perinatal asphyxia, acute illness, prematurity and congenital abnormality other than CHD.

Ages: 1 Day to 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: term newborns
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2014-04-30 (Actual); Study Completion 2014-05-31 (Actual)

PRIMARY OUTCOMES:
rSO2 | RSO2 values were obtained after 30 minute calm down period to enable stable recordings on each channel by averaging five minutes recorded values.
  regional tissue oxygenation assessed by NIRS

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided